CLINICAL TRIAL: NCT01138176
Title: Phase II Randomized Control Trial of Whole Body Cooling in Neonatal Encephalopathy Using Phase Changing Material
Brief Title: Whole Body Cooling Using Phase Changing Material
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Robertson, Nicola, M.D. (Individual)
Collaborators: Thayyil, Sudhin (Individual)
Responsible Party: Nicola Robertson, Reader in Translational Neonatal Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PCM09
Record Dates: First submitted 2010-06-02; First posted 2010-06-07 (Estimated); Last update posted 2010-06-07 (Estimated); Status verified 2010-06

CONDITIONS: Hypoxic Ischemic Encephalopathy
Keywords: Neonatal encephalopathy; Therapeutic hypothermia; Phase changing material; MR imaging
MeSH Terms: conditions — Hypoxia-Ischemia, Brain | interventions — Cool-Down Exercise; Hypothermia, Induced

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard care (No Intervention)
  Interventions: Procedure: Cooling
- Cooling (Experimental): Reduction of rectal temperature to 33.5 C for 72 hours
  Interventions: Procedure: Cooling

INTERVENTIONS:
Procedure: Cooling — Reduction of rectal temperature to 33.5 C
  Other Names: Therapeutic hypothermia; Whole body cooling

SUMMARY:
A prospective randomized control trial to examine safety and effectiveness of whole body cooling to a rectal temperature of 33.5 C using phase changing material in neonatal encephalopathy. Effectiveness will be defined by examining the stability of rectal temperature during cooling. Monitoring of vital signs, infection screen, blood counts, coagulation screen, liver and renal function tests, cranial US and MR imaging will be performed on recruited infants to evaluate safety of cooling. EEG will be performed on day 4 and hearing evaluation at discharge. Neurodevelopmental evaluation will be performed at 1 year of age.

DETAILED DESCRIPTION:
Meta-analyses of these trials show that therapeutic hypothermia increases survival with normal neurological function (pooled risk ratio of 1.53) with a number needed to treat of 8 (95% confidence interval (CI) 5 - 17) and in survivors reduces the rates of severe disability and cerebral palsy. Therapeutic hypothermia is now widely offered to moderately or severely asphyxiated infants in high-income countries.

The global burden of disease estimates indicate that perinatal asphyxia is a very significant problem in low and mid resourced settings. There are, however, several compelling reasons why the efficacy and safety data on therapeutic hypothermia from high-income countries cannot be extrapolated to neonatal units in transitional countries, such as India; in particular there is a lack of effective low tech servo controlled cooling equipments that can be used in these settings. This pilot phase II randomized control trial will examine the efficacy of phase changing material in providing satisfactory therapeutic hypothermia in neonatal encephalopathy, in a mid resource setting.

ELIGIBILITY:
Inclusion Criteria:

* Apgar score of <5 at 5 minutes or continued resuscitation at 5 minutes
* Neonatal encephalopathy

Exclusion Criteria:

* Imminent death
* Major congenital malformations
* Gestation <36 weeks
* Birthweight less than 1.8 kg

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Estimated)
Dates: Start 2009-07; Primary Completion 2011-01 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Stability of cooling | 72 hours
  Percentage of time for which rectal temperature is maintained between 33 to 34 C during the 72 hours of therapeutic hypothermia

SECONDARY OUTCOMES:
Brain tissue injury on MR imaging | 7 to 10 days
  Basal ganglia, white matter and cortical lesions scored from 0 to 3
Adverse neurodevelopment | 12 months
  severe neurodevelopmental impairment (defined as scores of <60 on neurological examination30 and/or a developmental score < 2SD (DASII) below the mean and/or GMFCS>II), microcephaly (head circumference <2 SD below mean), severe visual or hearing impairment
Mortality | 4 weeks
  Death until hospital discharge
EEG abnormality | 4 days
  Abnormal background activity
Sepsis | 1 week
  Blood or CSF culture positive sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Balraj Guhan, MD, Principal Investigator — Calicut Medical College
Locations (1):
- Calicut Medical College, Calicut, India

REFERENCES:
- See also: UCL Institute for Women's Health — http://www.instituteforwomenshealth.ucl.ac.uk/academic_research/neonatology